CLINICAL TRIAL: NCT00125645
Title: Global Left Ventricular Function After Acute Myocardial Infarction. Treatment With the Angiotensin 2-Receptor Blocker Irbesartan
Brief Title: Left Ventricular Function After Acute Myocardial Infarction (AMI). Treatment With Angiotensin 2-Receptor Blockade (GLOBAL-Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Kenneth Egstrup, Professor, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VF 20040053; 2612
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2007-04

CONDITIONS: Myocardial Infarction
Keywords: AMI; Left ventricular function; Myocardial performance index; Acute myocardial infarction (AMI)
MeSH Terms: conditions — Myocardial Infarction | interventions — Irbesartan

STUDY DESIGN:
Intervention Model Description: Comparison with EF

ARMS (1):
- Irbesartan (Experimental): Tablet Irbesartan 150 mg once daily
  Interventions: Drug: Irbesartan Oral Tablet

INTERVENTIONS:
Drug: Irbesartan Oral Tablet

SUMMARY:
The purpose of this study is to compare changes in global left ventricular (LV) function after 3 months of treatment with irbesartan compared with usual care in patients with acute myocardial infarction, a wall motion score >1.3 (EF>0.40) and signs of diastolic dysfunction. The hypothesis is that an angiotensin 2-receptor inhibitor will improve global left ventricular function.

DETAILED DESCRIPTION:
Study objectives:

Primary Objective:

To compare the change in global LV function assessed with myocardial performance index (MPI) after 3 months treatment with irbesartan compared to usual care in patients admitted to hospital with acute myocardial infarction, wall motion score index > 1.3 (LVEF > 0.40), and MPI > 0.55.

Secondary Objectives:

* To compare irbesartan added to an ACE-inhibitor compared to usual care in patients with AMI, WMSI <= 1.3 and MPI > 0.55;
* To compare LV diastolic function assessed by pulse wave and color M-mode Doppler echocardiography and left atrial size after treatment with irbesartan compared to usual care in AMI and

  * WMSI > 1.3 and MPI > 0.55; and
  * WMSI <= 1.3 and MPI > 0.55.
* To compare change in WMSI after treatment with irbesartan compared to usual care in patients with AMI and

  * WMSI > 1.3 and MPI > 0.55; and
  * WMSI <= 1.3 and MPI > 0.55.

Tertiary Objectives:

To assess the effects of irbesartan versus usual care on neurohormonal activation and glucose metabolism (optional).

Study Design:

A Danish multicenter randomized prospective trial with PROBE-design.

Study Drug:

Patients will be randomized to receive either: irbesartan 300 mg once daily or usual care.

Duration of Therapy:

Irbesartan 300 mg daily for 3 months after hospital discharge for acute myocardial infarction.

Patients should receive standard medical therapy including revascularisation as appropriate.

Expected Number of Patients:

200 patients with AMI, WMSI > 1.3 and MPI > 0.55 (100 patients in the irbesartan group and 100 in the usual care group). The patients will be included in the analysis of the primary endpoint. Further, approximately 100 patients with AMI, WMSI <= 1.3 and MPI > 0.55 treated with an ACE-inhibitor would be part of the secondary endpoints.

Main Inclusion Criteria:

* Patients admitted to hospital with clinical symptoms of acute myocardial infarction and/or electrocardiographic signs of AMI and a documented elevation in cardiac markers (troponin T or I) or elevation of cardiac enzymes (creatinine kinase MB).
* Myocardial performance index (MPI) > 0.55 determined by echocardiography prior to randomization.
* Be randomized within 7 days of AMI (in or out patient).
* Written informed consent

Main Exclusion Criteria:

* Age < 18 years.
* Any contraindications to angiotensin 2-receptor blocker.
* In patients with WMSI > 1.3 treatment with ACE-inhibitor or angiotensin 2-receptor blockers.
* In patients with WMSI <= 1.3 no initiated or planned treatment with an ACE-inhibitor. Treatment with an ACE-inhibitor must be started within 7 days.
* Pregnancy or women of childbearing potential who are not using an effective method of contraception.
* Other comorbid conditions that would influence the study.
* Currently receiving an experimental study-drug.

Study Medication:

Irbesartan 300 mg once daily which can be reduced to 150 mg at the discretion of the treating physician. With a dose less than 150 mg patients will be excluded from analysis.

Mode of Administration:

The drugs will be given unblinded, but with blinded assessment of the endpoints.

Evaluation Criteria:

Primary Outcome:

Change in MPI in patients with WMSI > 1.3 treated with either irbesartan or usual care.

Secondary Outcomes:

* Change in MPI in patients with WMSI <= 1.3 on an ACE-inhibitor treated with either irbesartan or usual care.
* Change in left ventricular diastolic function (pulse wave and color M-mode echocardiography and left atrial size) in patients with WMSI > 1.3 or <= 1.3.
* Change in LV systolic function (WMSI and LVEF) in patients with WMSI > 1.3 or WMSI <= 1.3.

Tertiary Outcomes:

Changes in neurohormonal activation and glucose metabolism (optional).

Definitions of Objectives:

Myocardial Performance Index:

MPI is calculated as the sum of the isovolumetric relaxation and contraction times divided by ejection time; this is measured from mitral inflow and left ventricular outflow recording obtained by pulse wave Doppler echocardiography.

LV Diastolic Function:

* Assessment of mitral inflow curve, E- and A-wave and deceleration time of the E-wave.
* Color M-mode:

Assessment of the flow propagation velocity.

* Left atrial size measured by single plane volume in a four chamber view.

Systolic Function:

* Wall motion score index: LV is divided into 16 segments which are scored based on myocardial thickening and endocardial excursion (3 = hyperkinesis, 2 = normokinesis, 1 = hypokinesis, 0 = akinesis and -1 = paradoxical motion). WMSI is calculated by dividing the sum of scores by the number of segments analyzed.
* LV ejection fraction is obtained by multiplying WMSI by 30.

Neurohormonal activation is assessed by pro-NT-BNP and glycemic control is assessed by an oral glucose tolerance test during hospitalisation and after 3 months in patients without known diabetes mellitus (optional).

Statistical Considerations:

Population Analyzed: All randomized patients will be in the study for the planned treatment period of 3 months, but only patients on >= 150 mg irbesartan will be analyzed according to the primary endpoint.

Sample Size Consideration: The primary study objective is to show that irbesartan will improve MPI more than usual care after 3 months treatment in patients with AMI, WMSI > 1.3 and MPI > 0.55.

Furthermore, patients with reduced LV function (WMSI <= 1.3) and with reduced global LV function (MPI > 0.55) will be included in the study and irbesartan will be added to an ACE-inhibitor compared to usual care. This patient will be included in the secondary objectives and therefore no sample size estimation has been performed. 100 patients are estimated to be enrolled in this study group and will be used for descriptive purposes.

It is assumed that MPI has a normal distribution in the study population and from previous populations of patients with AMI it is found, that MPIs have a mean value of 0.55 (SD 0.20) in patients with WMSI > 1.3; based on an estimated change in MPI of 20% in the irbesartan group a total of approximately 200 patients are needed for the study.

Duration of Treatment and Observations:

Treatment:

Patients will receive irbesartan 300 mg daily (at least 150 mg per day) for 3 months treatment.

The primary observation period will be 3 months corresponding to the treatment period, but vital status or hospitalisation will be noted after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented AMI; MPI > 0.55
* Randomized within 7 days of AMI
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Any contraindications to angiotensin 2-receptor blockade
* In patients with WMSI > 1.3 treatment with ACE-inhibitor or angiotensin 2-receptor blockers
* In patients with WMSI <= 1.3 no initiated or planned treatment with an ACE-inhibitor. Treatment with an ACE-inhibitor must be started within 7 days
* Pregnancy or women of childbearing potential who are not using an effective method of contraception
* Other comorbid conditions that could influence the study
* Currently receiving an experimental study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Asst. Professor, Study Chair — Department of Medical Research, SHF Svendborg
Locations (1):
- Kardiologisk Klinik, Centralsygehuset Esbjerg/Varde, Esbjerg, Denmark